CLINICAL TRIAL: NCT05762432
Title: A Pilot Open Label Prospective, Randomised, Study to Evaluate the Safety and Efficacy of Keneric Healthcare RTD Wound Dressing in the Treatment of Diabetic Foot Ulcers Compared to Standard of Care
Brief Title: Diabetic Foot Ulcer Research Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Community Pharmacology Services Ltd (Other)
Collaborators: Keneric Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPS22.007
Record Dates: First submitted 2023-02-17; First posted 2023-03-09 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot Ulcer Neuropathic; Diabetic Foot Ulcer Ischemic
Keywords: Diabetes; Foot Ulcer; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: Combination of normal standard of care and study device
Masking Description: Subjects will be randomised 1:1 to RTD Wound Dressing or standard of care dressing. Randomisation will be in blocks of four.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study Device (Experimental): This Arm of the study will receive the study device. Although the Study Device is not experimental as it is already CE marked and being used for it's intended purpose.
  Interventions: Device: Wound Dressing
- Standard of Care (Active Comparator): This arm of the study will use the NHS' existing standard of care device as is normally used in podiatry clinics.
  Interventions: Device: NHS Standard Dressing

INTERVENTIONS:
Device: Wound Dressing — RTD Wound Dressing that is being investigated
  Arms: Study Device
Device: NHS Standard Dressing — This is the standard dressing used by NHS staff when currently dealing with a diabetic foot ulcer
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to compare safety and performance of the study device to the current typical NHS standards of care device. The main outcomes it aims to achieve are:

Complete wound healing at 12 weeks (100% epithelialised)

% Reduction in wound area at 12 weeks

Participants will attend their NHS podiatry clinic appointment as normal and will be assigned either the study device or the current typical NHS standard of care device. Researchers will compare the study device group to the standard group to assess the outcomes mentioned previously.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to evaluate the safety and performance of the RTD Wound Dressing in the treatment of non-infected neuropathic, ischaemic, and neuro-ischaemic diabetic foot ulcers versus standard of care.

This clinical evaluation study will be performed under an open-label, comparative, design in the single health board of NHS Lanarkshire within 3 diabetic foot clinics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥18 years old with a diagnosis of type 1 or type 2 diabetes.
* New presentation for treatment of a neuropathic, ischaemic or neuro- ischaemic non- infected DFU
* Subjects must be able to follow verbal and written instructions in English
* Subjects must have full mental capacity and able to give written informed consent to participation in the trial including medical photography for the purposes of the clinical trial or clinical care.
* DFU is >10mm2 and <100mm2

Exclusion Criteria:

* Known allergy/hypersensitivity to any ingredient contained in the Keneric healthcare RTD Wound Dressing
* Participants who will have problems following the protocol, including the offloading system, provided as standard of care, to wear on a daily basis
* Suspected malignancy in the wound
* Critical limb ischaemia
* Pregnant or breastfeeding females
* Women of childbearing potential and not using a medically accepted form of contraception when sexually active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Completion of Wound Healing | 12 weeks
  100% epithelialised
Reduction in Wound Area | 12 weeks
  % reduction in size of Wound Area

SECONDARY OUTCOMES:
Wound Infection Rates | 12 weeks
  Rates at which the wound is infected
Dressing Changes | 12 weeks
  Number of dressing changes required per week and in total

CONTACTS AND LOCATIONS:
Overall Officials: Kaye McIntyre, MsC, Principal Investigator — NHS Lanarkshire
Locations (2):
- United Kingdom (2):
  - NHS Lanarkshire, Airdrie, North Lanarkshire
  - NHS Lothian, Livingston, West Lothian

IPD SHARING:
Plan to Share IPD: No
No data will be shared.